CLINICAL TRIAL: NCT02174328
Title: Prevention of Preeclampsia With Aspirin Administered From the Beginning of Pregnancy in Recipients of Donated Oocytes.
Brief Title: Prevention of Preeclampsia With Aspirin in Recipients of Donated Oocytes.
Acronym: PROVAS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Halted prematurely due to low recruitment rate.
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PrOvAS001
Record Dates: First submitted 2013-09-11; First posted 2014-06-25 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Pre-Eclampsia
Keywords: See incidence of Pre-Eclampsia in acetylsalicylic acid group; See incidence of Pre-Eclampsia in placebo group
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetylsalicylic acid (Experimental): This group will receive 1 tablet of acetylsalicylic acid (100 mg) orally daily from 5-10 weeks gestation until the end of gestation, about week 36
  Interventions: Drug: Acetylsalicylic acid
- Placebo (Placebo Comparator): This group will receive 1 tablet of placebo orally each day from 5-10 weeks gestation until the end of gestation, about week 36
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid — Acetylsalicylic acid once a day until 36 week
  Other Names: ADIRO 100
  Arms: acetylsalicylic acid
Drug: Placebo — Placebo once a day until 36 week
  Other Names: Not active drug
  Arms: Placebo

SUMMARY:
The main objective of this trial is to study the occurrence of preeclampsia in recipients of donated oocytes receiving aspirin at an early stage during pregnancy and to compare the results with those obtained in patients receiving placebo.

DETAILED DESCRIPTION:
Various markers have been proposed for the early diagnosis of preeclampsia: determination of mean arterial pressure; presence of multiple risk factors of preeclampsia; biochemical, ultrasound, and angiogenic markers; uterine artery Doppler, etc. These are used to determinate which patients have an increased risk of developing preeclampsia during gestation, and therefore carry out closer monitoring of pregnancy in this population. In addition, these markers can also identify patients at increased risk of developing other problems such as IUGR or preterm labor.

For nearly 30 years, there have been multiple studies trying to demonstrate that aspirin prevents the onset of preeclampsia with inconclusive results. However, recent studies in which aspirin was administered at an early stage (before 16 weeks of gestation) in patients at high risk of complications, have demonstrated a decrease in the incidence of this entity. Thus, administration of aspirin to patients at high risk (patients classified with a high risk of complications during pregnancy, based on markers mentioned above) seems to be useful in preventing onset of preeclampsia, IUGR and other complications, whenever it is administered at an early stage, as shown by several studies carried out so far.

The incidence of preeclampsia, IUGR and other complications of pregnancy is increased in patients undergoing treatment for ovulation induction, being much higher in recipients of donated oocytes. It appears that this increase may be explained by immunological processes. The focus lies on the interaction between HLA-C fetal antigen with the maternal natural killer cells. We postulate, therefore, that the administration of aspirin in recipients of donated oocytes at an early stage of pregnancy, may also reduce the incidence of preeclampsia in this group of patients.

Moreover, it has been observed that patients with preeclampsia exhibit lower levels of VEGF, PlGF and PAPP-A (factors involved in placental angiogenesis) and that this is accompanied by an increase in the sFlt1 (a potent PIGF and VEGF antagonist).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years.
* Recipients of donated oocytes.
* Pregnant women.
* Single or twin gestations.
* Patients who accept the conditions of the study by signing the appropriate informed consent.

Exclusion Criteria:

* Known allergy to acetylsalicylic acid .
* Personal history of peptic ulcer.
* Triplets.
* Use of prostaglandin inhibitors within 10 days prior to baseline.
* Personal history of chronic kidney, thyroid, liver or heart disease.
* Psychiatric or cognitive pathology that prevents understanding of the conditions of informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Occurrence of preeclampsia. | Up to 42 weeks
  The main objective is to study the occurrence of preeclampsia in recipients of donated oocytes receiving aspirin at an early stage during pregnancy, and to compare the results with those obtained in patients receiving placebo.

SECONDARY OUTCOMES:
Other complications | Up to 42 weeks
  Determine the development of gestational hypertension, severe preeclampsia, IUGR, and preterm delivery in this group of patients.

OTHER OUTCOMES:
Inflammatory mediators involved in angiogenesis. | Up to 42 weeks
  Another objective is to determine if aspirin, through blockade of cyclooxygenase-2, could act in addition to reducing the synthesis of thromboxane 2, altering or diminishing the formation of various inflammatory mediators involved in angiogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Perales, PhD, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Obstetrics Unit of La Fe University and Politechnic Hospital, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebrashy A, Ibrahim M, Marzook A, Yousef D. Usefulness of aspirin therapy in high-risk pregnant women with abnormal uterine artery Doppler ultrasound at 14-16 weeks pregnancy: randomized controlled clinical trial. Croat Med J. 2005 Oct;46(5):826-31. PMID 16158479
- [Background] ACOG Committee on Practice Bulletins--Obstetrics. ACOG practice bulletin. Diagnosis and management of preeclampsia and eclampsia. Number 33, January 2002. Obstet Gynecol. 2002 Jan;99(1):159-67. doi: 10.1016/s0029-7844(01)01747-1. PMID 16175681
- [Background] Akolekar R, de Cruz J, Foidart JM, Munaut C, Nicolaides KH. Maternal plasma soluble fms-like tyrosine kinase-1 and free vascular endothelial growth factor at 11 to 13 weeks of gestation in preeclampsia. Prenat Diagn. 2010 Mar;30(3):191-7. doi: 10.1002/pd.2433. PMID 20101671
- [Background] Akolekar R, Syngelaki A, Sarquis R, Zvanca M, Nicolaides KH. Prediction of early, intermediate and late pre-eclampsia from maternal factors, biophysical and biochemical markers at 11-13 weeks. Prenat Diagn. 2011 Jan;31(1):66-74. doi: 10.1002/pd.2660. PMID 21210481
- [Background] Akolekar R, Zaragoza E, Poon LC, Pepes S, Nicolaides KH. Maternal serum placental growth factor at 11 + 0 to 13 + 6 weeks of gestation in the prediction of pre-eclampsia. Ultrasound Obstet Gynecol. 2008 Nov;32(6):732-9. doi: 10.1002/uog.6244. PMID 18956425
- [Background] Audibert F, Boucoiran I, An N, Aleksandrov N, Delvin E, Bujold E, Rey E. Screening for preeclampsia using first-trimester serum markers and uterine artery Doppler in nulliparous women. Am J Obstet Gynecol. 2010 Oct;203(4):383.e1-8. doi: 10.1016/j.ajog.2010.06.014. Epub 2010 Aug 5. PMID 20691410
- [Background] Brosens I, Pijnenborg R, Vercruysse L, Romero R. The "Great Obstetrical Syndromes" are associated with disorders of deep placentation. Am J Obstet Gynecol. 2011 Mar;204(3):193-201. doi: 10.1016/j.ajog.2010.08.009. Epub 2010 Nov 20. PMID 21094932
- [Background] Brown MA, Lindheimer MD, de Swiet M, Van Assche A, Moutquin JM. The classification and diagnosis of the hypertensive disorders of pregnancy: statement from the International Society for the Study of Hypertension in Pregnancy (ISSHP). Hypertens Pregnancy. 2001;20(1):IX-XIV. doi: 10.1081/PRG-100104165. No abstract available. PMID 12044323
- [Background] Bujold E, Roberge S, Lacasse Y, Bureau M, Audibert F, Marcoux S, Forest JC, Giguere Y. Prevention of preeclampsia and intrauterine growth restriction with aspirin started in early pregnancy: a meta-analysis. Obstet Gynecol. 2010 Aug;116(2 Pt 1):402-414. doi: 10.1097/AOG.0b013e3181e9322a. PMID 20664402
- [Background] Imperiale TF, Petrulis AS. A meta-analysis of low-dose aspirin for the prevention of pregnancy-induced hypertensive disease. JAMA. 1991 Jul 10;266(2):260-4. PMID 1829118
- [Background] Keegan DA, Krey LC, Chang HC, Noyes N. Increased risk of pregnancy-induced hypertension in young recipients of donated oocytes. Fertil Steril. 2007 Apr;87(4):776-81. doi: 10.1016/j.fertnstert.2006.08.105. Epub 2007 Jan 29. PMID 17258714
- [Background] Klatsky PC, Delaney SS, Caughey AB, Tran ND, Schattman GL, Rosenwaks Z. The role of embryonic origin in preeclampsia: a comparison of autologous in vitro fertilization and ovum donor pregnancies. Obstet Gynecol. 2010 Dec;116(6):1387-1392. doi: 10.1097/AOG.0b013e3181fb8e59. PMID 21099607
- [Background] Levine RJ, Lam C, Qian C, Yu KF, Maynard SE, Sachs BP, Sibai BM, Epstein FH, Romero R, Thadhani R, Karumanchi SA; CPEP Study Group. Soluble endoglin and other circulating antiangiogenic factors in preeclampsia. N Engl J Med. 2006 Sep 7;355(10):992-1005. doi: 10.1056/NEJMoa055352. PMID 16957146
- [Background] Le Ray C, Scherier S, Anselem O, Marszalek A, Tsatsaris V, Cabrol D, Goffinet F. Association between oocyte donation and maternal and perinatal outcomes in women aged 43 years or older. Hum Reprod. 2012 Mar;27(3):896-901. doi: 10.1093/humrep/der469. Epub 2012 Jan 16. PMID 22252087
- [Background] Lambers MJ, Groeneveld E, Hoozemans DA, Schats R, Homburg R, Lambalk CB, Hompes PG. Lower incidence of hypertensive complications during pregnancy in patients treated with low-dose aspirin during in vitro fertilization and early pregnancy. Hum Reprod. 2009 Oct;24(10):2447-50. doi: 10.1093/humrep/dep245. Epub 2009 Jul 16. PMID 19608566
- [Background] Nicolaides KH. A model for a new pyramid of prenatal care based on the 11 to 13 weeks' assessment. Prenat Diagn. 2011 Jan;31(1):3-6. doi: 10.1002/pd.2685. No abstract available. PMID 21210474
- [Background] Pecks U, Maass N, Neulen J. Oocyte donation: a risk factor for pregnancy-induced hypertension: a meta-analysis and case series. Dtsch Arztebl Int. 2011 Jan;108(3):23-31. doi: 10.3238/arztebl.2011.0023. Epub 2011 Jan 21. PMID 21285999
- [Background] Poon LC, Akolekar R, Lachmann R, Beta J, Nicolaides KH. Hypertensive disorders in pregnancy: screening by biophysical and biochemical markers at 11-13 weeks. Ultrasound Obstet Gynecol. 2010 Jun;35(6):662-70. doi: 10.1002/uog.7628. PMID 20232288
- [Background] Ruano R, Fontes RS, Zugaib M. Prevention of preeclampsia with low-dose aspirin -- a systematic review and meta-analysis of the main randomized controlled trials. Clinics (Sao Paulo). 2005 Oct;60(5):407-14. doi: 10.1590/s1807-59322005000500010. Epub 2005 Oct 24. PMID 16254678
- [Background] Salha O, Sharma V, Dada T, Nugent D, Rutherford AJ, Tomlinson AJ, Philips S, Allgar V, Walker JJ. The influence of donated gametes on the incidence of hypertensive disorders of pregnancy. Hum Reprod. 1999 Sep;14(9):2268-73. doi: 10.1093/humrep/14.9.2268. PMID 10469693
- [Background] Simhan HN, Caritis SN. Prevention of preterm delivery. N Engl J Med. 2007 Aug 2;357(5):477-87. doi: 10.1056/NEJMra050435. No abstract available. PMID 17671256
- [Background] Smith GC, Stenhouse EJ, Crossley JA, Aitken DA, Cameron AD, Connor JM. Early pregnancy levels of pregnancy-associated plasma protein a and the risk of intrauterine growth restriction, premature birth, preeclampsia, and stillbirth. J Clin Endocrinol Metab. 2002 Apr;87(4):1762-7. doi: 10.1210/jcem.87.4.8430. PMID 11932314
- [Background] Soderstrom-Anttila V. Pregnancy and child outcome after oocyte donation. Hum Reprod Update. 2001 Jan-Feb;7(1):28-32. doi: 10.1093/humupd/7.1.28. PMID 11212070
- [Background] Soderstrom-Anttila V, Tiitinen A, Foudila T, Hovatta O. Obstetric and perinatal outcome after oocyte donation: comparison with in-vitro fertilization pregnancies. Hum Reprod. 1998 Feb;13(2):483-90. doi: 10.1093/humrep/13.2.483. PMID 9557862
- [Background] Groeneveld E, Lambers MJ, Lambalk CB, Broeze KA, Haapsamo M, de Sutter P, Schoot BC, Schats R, Mol BW, Hompes PG. Preconceptional low-dose aspirin for the prevention of hypertensive pregnancy complications and preterm delivery after IVF: a meta-analysis with individual patient data. Hum Reprod. 2013 Jun;28(6):1480-8. doi: 10.1093/humrep/det022. Epub 2013 Mar 25. PMID 23528915